CLINICAL TRIAL: NCT06459960
Title: Effect of a Tailor-made Hydrotherapy on Physical Functions in Patients After Unilateral Unicompartmental Knee Arthroplasty
Brief Title: Effect of Hydrotherapy After Unilateral UKA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Ho Ki Wai, Clinical Professional Consultant, Chinese University of Hong Kong
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020.586
Record Dates: First submitted 2024-06-11; First posted 2024-06-14 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Osteoarthritis, Knee
Keywords: unicompartmental knee arthroplasty; hydrotherapy; physical function
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Hydrotherapy; Congresses as Topic

STUDY DESIGN:
Intervention Model Description: Patients were divided into 1) hydrotherapy group (Hydrotherapy) or 2) convention group (Convention)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hydrotherapy (Experimental): Patients practised the rehabilitation exercises in a heated pool (32°C). Exercises included: 1) Knee mobilization exercises, 2) Muscle stretching exercises, 3) Muscle strengthening exercises, such as wall slide, leg press with life ring, and lunges, 4) Balance and functional training - Single-leg standing, tandem walking, heel walking and tip-toe walking, and 5) Balance functional training - Cycling in water, fast walking and running (for patients in Hydrotherapy group only).
  Patients practised once a week for a total of four weeks, complimentary to conventional physiotherapy rehabilitation (8 weeks). Total number of weeks is 8+4 weeks = 12 weeks.
  Interventions: Genetic: Hydrotherapy
- Convention (Active Comparator): The conventional physiotherapy rehabilitation programme included: 1) knee mobilization exercises, such as static bike and heel sliding board, 2) Muscle stretching exercises of hamstrings and calf, 3) Muscle strengthening exercises, such as adding cuff weights for quadriceps strengthening and wall slide with gym ball, and 4) Balance and functional training, such as stepping or single-leg standing on soft foam, stepping exercises on various heights of steps.
  Patients practised twice a week for a total of 8 weeks.
  Interventions: Genetic: Convention

INTERVENTIONS:
Genetic: Hydrotherapy — Heated pool (32°C); Convention rehabilitation + Hydrotherapy
  Arms: Hydrotherapy
Genetic: Convention — Convention rehabilitation only
  Arms: Convention

SUMMARY:
Osteoarthritis (OA) is a progressive disease of the synovial joints that causes joint pain and limitation of function resulting in considerable morbidity and impairment of quality of life. Knee OA is the most common type of OA, and symptomatic knee OA is highly prevalent among people aged over 50 years. With the increasing aging population, worldwide prevalence of knee OA is expected to be rising. The goals of treatment are to reduce pain, maintain or improve joint mobility, minimize functional impairment and improve quality of life. When conservative management, which includes structured land-based exercise programs, aquatic exercise, education and appropriate analgesic medications, fails, surgical approach can be considered. Unicompartmental knee arthroplasty (UKA) has become an alternative to TKA in cases of end-stage OA that are limited to a single compartment. Patients who underwent UKA have a quicker recovery, lower risk of complications, and improved range of motion. Physiotherapy rehabilitation is an integral part of good knee arthroplasty outcome. Conventional post-operative physiotherapy rehabilitation, which includes range of motion exercises, muscle strengthening exercises, balance and gait training, have been shown to have improvement in range of motion, muscle strength and functional outcome measures of patients. Recently, hydrotherapy is gaining its popularity as being incorporated into one of the components in the rehabilitation after knee arthroplasty. Studies reported that hydrotherapy could decrease pain, and improved physical function, strength and quality of life for patients after total hip or knee arthroplasty. However, there are no studies to investigate the effect of hydrotherapy on patients after UKA. With the increasing popularity of UKA as a surgical alternative in patients with end-stage single-compartmental OA, it is worth investigating the effects of hydrotherapy on the clinical outcomes of patients following UKA.

DETAILED DESCRIPTION:
Osteoarthritis (OA) of the knee is one of the most common chronic degenerative joint diseases, primarily affecting the ageing population, limiting joint movement and causing disability because of pain and stiffness. Prevalence of radiologic knee OA increased in proportion to age, reaching 64.1% for those who were aged 60 and over, and had a higher prevalence in females than males. OA is a progressive joint disorder, characterized by progressive softening and disintegration of articular cartilage, growth of osteophytes and fibrosis of joint capsule. Clinical presentations vary from asymptomatic despite the presence of radiological evidence, to progressively evolving symptoms and eventually severely disabling joints. Knee OA is the most common type of OA, affecting patello-femoral joint and/or medial tibio- femoral joint. Symptoms of knee OA include joint pain, knee effusion, quadriceps muscle weakness and wasting, giving way, and knee deformities such as fixed flexion contractures and varus knees. These can lead to functional limitations, resulting in substantial morbidity and impaired quality of life. The Global Burden of Diseases studies reported that OA was the leading cause of lower extremity disability in elderly, with hip and knee OA accounting for 1.12% of years lived with disability. OA has been reported to be ranked the seventh leading cause of global years lived with disability. Moreover, knee OA leads to substantial medical expenses and economic burden. Patients suffering from knee OA flock to general practitioners and orthopaedic specialists for analgesic medications and injections, or physiotherapists for exercise consultations, or orthopaedic surgeons for surgery. These reactions subsequently become burden to healthcare systems and expenses leading to healthcare dilemmas.

The ever-aging population proved to be one of the strongest predictors of OA, particularly in patients with age 50 years and higher. Studies reported that there was a high prevalence of symptomatic knee OA among people aged over 50 years, affecting more than 250 million people worldwide. With the growing aging population, worldwide prevalence of knee OA is expected to be rising. Therefore, knee OA is gaining attention from our society, policy makers and medical professionals on its management, aiming at holistic, cost-effective and evidence-based care approach. Management of knee OA can be classified into conservative and surgical approaches, aiming at reducing pain, maintaining or improving joint mobility, minimizing functional impairment and improving quality of life. For conservative approach, a combination of non-pharmacological and pharmacological modalities, which include structured land-based exercise programs, aquatic exercise, education and appropriate analgesic medications, are recommended and supported by evidence.

Surgery is the subsequent approach after failure in conservative management. Total knee arthroplasty (TKA) has been the dominating surgery for patients who suffer from severe end- stage symptomatic OA but fail to respond to conservative management and have significantly impaired function and quality of life. Recently, unicompartmental knee arthroplasty (UKA) has become an alternative to TKA for patients with end-stage knee OA.

Patients after UKA reported quicker recovery period, lower risk of complications and better range of motion if the knee. Our group investigated the correlation between femoral and tibial component axial rotational alignment and functional outcomes in 83 Oxford UKA from in 67 patients with isolated medial or lateral compartment knee osteoarthritis. We found that femoral component axial rotation between 2° and 6° external rotation, and tibial component axial rotation between 1° and 8° external rotation correlated with significantly better functional scores, with the highest functional scores observed at 3°-4° external rotation for femoral component, and 4°-5° external rotation for tibial component.

After knee arthroplasty, physiotherapy rehabilitation is a part of non-invasive treatments leading to a successful outcome after surgery. Conventional post-operative physiotherapy, including exercises aiming at improving range of motion, muscle strengthening, body balance and gait training, showed to have improvement in range of motion and muscle strength of knee. An European review on exercises after knee arthroplasty reported improvements in various functional outcome measures such as Western Ontario and McMaster Universities Arthritis Index (WOMAC), Medical Outcome Study Short Form-36 (SF-36), Oxford Knee Score, American Knee Society Score, Lower Extremity Functional Scale and Iowa Lower Extremity Scale.

Recently, hydrotherapy is gaining popularity on its use being an important component in rehabilitation programme after knee arthroplasty. Hydrotherapy is the external or internal use of water in any of its forms (water (liquid), ice (solid), steam (gas)) for health promotion or treatment of various diseases with various temperatures, pressure, duration, and site. In clinical settings, patients exercise in a temperature-controlled water pool led by a physiotherapist. Exercising in water has a long history of beneficial therapeutic effect to promote healing in certain medical conditions. Hydrotherapy has been widely used in various musculoskeletal and neurologic conditions, from paediatric to geriatric population. Patients exercising in a hydrotherapy pool could perform better than on land and let patients who could not perform the same exercise on land work out under water. Benefits of warm-bathing hydrotherapy include relieving pain and muscle spasm through warmth, reducing loading of joints through buoyancy, decreasing oedema through pressure from immersion, and producing resistance to movement through turbulence and hydrostatic pressure. Studies proved that hydrotherapy could decrease pain, and improve physical functions, muscle strength and quality of life in patients after total hip or knee arthroplasty.

Given the benefits of hydrotherapy on patients who underwent joint replacement, there is no study investigating the effect of hydrotherapy on patients after UKA. With the increasing popularity of UKA as a surgical alternative to TKA for patients with end stage single-compartmental knee OA, it is worth investigating the effects of hydrotherapy on the clinical outcomes of patients following UKA. Results can guide further discussions on whether hydrotherapy should be incorporated into the post-joint replacement surgery physiotherapy rehabilitation in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients who aged 18 or above, and underwent primary unilateral UKA , with the Oxford model, at the Department of Orthopaedics and Traumatology of the Alice Ho Miu Ling Nethersole Hospital (AHNH) in year 2018 and 2019 were included.

Exclusion Criteria:

* Patients who had post operative complications, underwent revision or robotic assisted surgery or bilateral knee arthro plasty, defaulted follow up, received post operative physiotherapy rehabilitation which was not at the Physiotherapy Department of AHNH, had cognitive impairment, or were unsuitable for exercise training, were excluded in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
Knee Society Function Score (KFS) | Baseline (Before surgery), Post-op 6 months, Post-op 1 year
  KFS is widely adopted as an outcome measure in knee arthroplasty related research. KFS assesses the patient's walking distance, stairs performance and the use of walking aid. The full mark is 100, with higher marks indicating better knee function and vice versa

SECONDARY OUTCOMES:
Self-reported walking tolerance (minutes) | Post-op first session and Post-op last session of rehabilitation programme; 12 weeks apart for Hydrotherapy group and 8 weeks apart for Convention group.
  Self-reported walking tolerance is a self-reported walking tolerance test to test the maximum time (in minutes) to tolerate walking before taking a rest.
Timed Up and Go Test (TUGT) (seconds) | Post-op first session and Post-op last session of rehabilitation programme; 12 weeks apart for Hydrotherapy group and 8 weeks apart for Convention group.
  TUGT measures the time required for the patient to rise from an armchair under standardized seat height, follow by walking for three meters, then return to sitting on the same chair.
30-second Chair Stand Test (30CST) (repetitions) | Post-op first session and Post-op last session of rehabilitation programme; 12 weeks apart for Hydrotherapy group and 8 weeks apart for Convention group.
  30CST measures the number of cycles or repetitions of continuous standing up and sitting down from a designated chair in 30 seconds. The test begins with the subject seated. The subject is then asked to rise from chair with arms folded across chest after command at the preferred speed.
Numeric pain rating scale (NPRS) | Post-op first session, Post-op 4 weeks, and 3) Post-op last session of rehabilitation programme; 12 weeks apart for Hydrotherapy group and 8 weeks apart for Convention group
  NPRS has been routinely applied to let patients rate the pain level on a defined scale. NPRS is a single 11-point numeric scale ranging between 0 and 10, with 0 representing "no pain" and 10 representing the pain extreme.
Passive range of motion - Flexion and Extension | Post-op first session, Post-op 4 weeks, and 3) Post-op last session of rehabilitation programme; 12 weeks apart for Hydrotherapy group and 8 weeks apart for Convention group.
  Passive ROM is the ability of a joint to be moved through its normal arc of motion while relaxed and the motion was performed by an outside force, for example, the therapist's hand, the client's opposite hand, or gravity. Passive ROM allows the assessor to focus on the quality of the joint structure and ligaments.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Ki-Wai Ho, FRCSEDOrtho, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Alice Ho Miu Ling Nethersole Hospital, Tai Po, N.T., Hong Kong

IPD SHARING:
Plan to Share IPD: No
Share among Study PI and research assistants within the facility only.

REFERENCES:
- [Derived] Chau WW, Lau MY, Choi TL, Lam GY, Ong MT, Ho KK. Effect of a tailor-made hydrotherapy on physical functions in patients after unilateral unicompartmental knee arthroplasty-A feasibility study. Arthroplasty. 2025 Feb 5;7(1):9. doi: 10.1186/s42836-024-00291-x. PMID 39905574